CLINICAL TRIAL: NCT01313455
Title: Adrenal Hyperplasia Among Young Patients With Polycystic Ovarian Syndrome
Brief Title: Adrenal Hyperplasia Among Young People With PCOS
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 110119; 11-CH-0119
Record Dates: First submitted 2011-03-10; First posted 2011-03-11 (Estimated); Last update posted 2019-05-31 (Actual); Status verified 2017-10-24

CONDITIONS: Adrenal Hyperplasia; Polycystic Ovarian Syndrome; Oligomenorrhea; Obesity; Hyperandrogenism
Keywords: Oligomenorrhea; Adrenal Hyperplasia; Obesity; Hyperandrogenism; Polycystic Ovarian Syndrome; PCOS; Polycystic Ovary; Healthy Volunteer; HV
MeSH Terms: conditions — Adrenal Hyperplasia, Congenital; Polycystic Ovary Syndrome; Oligomenorrhea; Obesity; Hyperandrogenism

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- Polycystic ovarian syndrome (PCOS) is a group of disorders related to problems with the secretion of certain hormones, which can lead to reproductive and other issues in women. Frequent complications of PCOS include irregular menstruation, development of ovarian cysts, and insulin resistance. The adrenal glands, which sit on top of the kidney, are involved in the production of certain hormones and the regulation of steroid levels in the blood, and may be affected in women with PCOS. Researchers are interested in studying possible connections between the adrenal glands and PCOS in young women who have been diagnosed with PCOS and healthy volunteers with normal menstrual function.

Objectives:

- To investigate possible connections between adrenal gland steroid hormone secretion and polycystic ovarian syndrome.

Eligibility:

* Women between 16 and 29 years of age who have been diagnosed with PCOS, or who are healthy volunteers with normal menstrual function.
* Participants must be willing to discontinue the use of oral contraceptives or any other medications that alter steroid hormone production for at least 1 month before the start of the study.

Design:

* Participants will be screened with a physical examination, medical history, and blood and urine tests. All participants will also have a pelvic (ovarian) ultrasound.
* All participants will be admitted to the hospital for a 1-week testing period, which will involve the following tests:
* Regular blood draws for two 2-hour periods (late evening and early morning) to measure hormone levels
* Fasting blood draws with a dose of corticotropin to test the body's adrenal function
* Hormone level measurement following regular doses of dexamethasone (a drug that controls the function of the adrenal gland)
* Daily urine collection for 6 days.
* Other studies, such as imaging studies of the adrenal glands, may be conducted as required by the study researchers.

DETAILED DESCRIPTION:
Polycystic ovarian syndrome (PCOS) is a heterogeneous group of disorders presenting with hyperandrogenism in adolescents and young women. The etiology of this condition remains unknown, despite its many identified links to insulin resistance, hypertension and metabolic syndrome, as well as its potential connection to the various forms of congenital adrenal hyperplasia (CAH).

The adrenal glands are the only source in the body of adrenocortical steroids. In normal physiology, the pituitary hormone ACTH regulates the secretion of glucocorticoids, while the secretion of mineralocorticoids is controlled by the renin-angiotensin system. In addition to these two steroids, the adrenal gland secretes lesser amounts of intermediate metabolites of these steroids, as well as the sex-steroids DHEA, DHEAS, androstenedione, testosterone, estrogen, and estrone. Dysregulated secretion of any of these hormones can be caused by the development of hyperplasia of the adrenocortical tissue, which may be mild and lead to specific clinical syndromes depending on the identity of the secreted hormones. Bilateral adrenocortical hyperplasia (BAH) is now an increasingly diagnosed cause of adrenal dysfunction.

We propose that there is a subgroup of patients with PCOS who actually have non-CAH primary forms of BAH. To investigate this possibility, we propose to study the hypothalamic-pituitary-adrenal axis (HPAA) over the next 2 years in 120 young girls and women (ages 16 to 25 years) that we will compare to 30 age- and race-matched normal females. Patients will be recruited primarily (although not exclusively) from a busy New York City clinic run by the Pediatric Endocrine Division at the Infants and Children's Hospital of Brooklyn at Maimonides and SUNY Downstate. All patients will undergo standard testing of the HPAA including oral low- and high-dose dexamethasone (DEX)-suppression testing (Liddle s test). Paradoxical rise of cortisol and/or other steroid metabolites in response to DEX is considered a sensitive test for the diagnosis of BAH. Patients with such responses will be molecularly investigated for the known causes of BAH (GNAS, PRKAR1A, PDE11A, PDE8B and other mutations).

The first goal of this study is to identify any possible contributions of the BAH phenotypes and genotypes to the pathophysiology of PCOS, a yet unknown factor in the etiology of this multifaceted disorder. The second goal is to perform a comparative analysis of the expression of large sets of genes in cells of these patients using gene arrays and other genetic analyses. This study will generate important information about the molecular pathways that are affected in this subgroup of patients with PCOS. Thirdly, this study will also allow for the collection of DNA from affected and non-affected relatives of the patients to perform genetic studies and identify causative genetic defects. Finally, the study is expected to lead to new diagnostic and therapeutic methods for at least certain forms of PCOS.

ELIGIBILITY:
* INCLUSION CRITERIA FOR PATIENTS:

Women 16-24 years old with PCOS defined as biochemical hyperandrogenism with associated findings of either menstrual irregularity and /or polycystic ovaries on ultrasound; hyperandrogenism defined as elevation of any of the following androgens: free testosterone, total testosterone, DHEAS, DHEA, 17 0H progesterone, androstenedione, 17OH pregnenolone; a polycystic ovary on ultrasound should either have 12 follicles measuring 2-9 mm in diameter, or have an increased ovarian volume of 10 CC or greater; menstrual irregularity defined as: Amenorrhea refers to absence of bleeding for at least three usual cycle lengths; oligomenorrhea refers to bleeding that occurs at an interval greater than 35 days.

We would like patients to have oligomenorrhea for at least six usual cycle lengths. Patients have to be off oral contraceptive pills or any other medications that alter steroidogenesis for at least one month prior to participating in the study

INCLUSION CRITERIA FOR CONTROLS:

Women 18-25 years old with normal menstrual function; they have to be off oral contraceptive pills or any other medications that alter steroidogenesis for at least one month prior to participating in the study.

EXCLUSION CRITERIA FOR PATIENTS:

Patients who have hyperandrogenism due to 21 hydroxylase deficiency non- classic adrenal hyperplasia androgen secreting neoplasms

Women with known or suspected androgenic/anabolic drug use

Women with severe insulin resistance-acanthosis nigricans syndrome; Fasting insulin levels are obtained to rule out syndromes of severe insulin resistance and hyperandrogenism; if insulin is above 80 mU/mL in the fasting state, and/or >300 mU/mL following a 2- or 3-hour oral glucose tolerance test (obtained elsewhere), patients are not eligible.

Women with thyroid dysfunction, hyperprolactinemia, (defined as prolactin level greater than or equal to 3 times the upper reference limit), less than 2 years post menarche, and patients on medications that alter steroidogenesis such as oral contraceptive pills, for less than a month prior to the date of inclusion in the study. (see above: patients have to be off oral contraceptive pills or any other medications that alter steroidogenesis for at least one month prior to participating in the study)

Women with prior history of pregnancy.

EXCLUSION CRITERIA FOR CONTROLS:

Young women with hyperandrogenemia, hirsutism or known adrenal tumors or other endocrine diseases, patients on multiple medications, known insulin resistance, or any other chronic or acute illness are not eligible as controls for this study.

Ages: 16 Years to 29 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 96 (Actual)
Dates: Start 2011-03-10; Study Completion 2017-10-24

CONTACTS AND LOCATIONS:
Overall Officials: Maya B Lodish, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Rosenfield RL. What every physician should know about polycystic ovary syndrome. Dermatol Ther. 2008 Sep-Oct;21(5):354-61. doi: 10.1111/j.1529-8019.2008.00217.x. PMID 18844713
- [Background] Karch S, Manzambi ZA, Salaun JJ. Field trials with Vectolex (Bacillus sphaericus) and Vectobac (Bacillus thuringiensis (H-14)) against Anopheles gambiae and Culex quinquefasciatus breeding in Zaire. J Am Mosq Control Assoc. 1991 Jun;7(2):176-9. PMID 1895075
- [Background] Krone N, Arlt W. Genetics of congenital adrenal hyperplasia. Best Pract Res Clin Endocrinol Metab. 2009 Apr;23(2):181-92. doi: 10.1016/j.beem.2008.10.014. PMID 19500762
- [Derived] Gourgari E, Lodish M, Keil M, Sinaii N, Turkbey E, Lyssikatos C, Nesterova M, de la Luz Sierra M, Xekouki P, Khurana D, Ten S, Dobs A, Stratakis CA. Bilateral Adrenal Hyperplasia as a Possible Mechanism for Hyperandrogenism in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2016 Sep;101(9):3353-60. doi: 10.1210/jc.2015-4019. Epub 2016 Jun 23. PMID 27336356